CLINICAL TRIAL: NCT05823168
Title: The Predictive Role of Seizures and Anitiepileptic Therapy on Rehabilitation Course of Traumatic Brain Injury
Brief Title: Seizures and Traumatic Brain Injury Rehabilitation
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Other Study IDs: 2503
Record Dates: First submitted 2023-03-06; First posted 2023-04-21 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Seizures; Traumatic Brain Injury
Keywords: rehabilitation; outcome; prophylaptic therapy
MeSH Terms: conditions — Seizures; Brain Injuries, Traumatic | interventions — Anticonvulsants

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with seizures: patients with traumatic brain injury
  Interventions: Drug: Antiepileptic Drug
- patients without seizures: patients with traumatic brain injury
  Interventions: Drug: Antiepileptic Drug

INTERVENTIONS:
Drug: Antiepileptic Drug — we osberve the efficacy of antiepileptic drungs on preventing seizures and their impact on rehabilitation outcome
  Other Names: antiepileptic prophylactic therapy

SUMMARY:
post-traumatic seizures (PTS) are a common and debilitating complication of traumatic brain injury (TBI) and could have harmful impact on patient disabilty and rehabilitation outcome.

In this multicentric prospective observational study we aimed to evaluate the role on functional outcome of patients admitted to neurorehabilitation unit afther traumatic brain injury of:

* newly occurring seizures
* prescription of antiepileptic prophylactic therapy

The inclusion criteria were the following: 1) age ≥ 18; 2) diagnosis of TBI on presentation; 3) admission to a hospital emergency department within 24 h of injury; 4) admission within one month from the injury to the rehabilitation unit to continue clinical care and rehabilitation program; 5) up to 6 months of observation in rehabilitation setting.

Were collected the following variables: gender, medical history, age at occurrence of injury, injury characteristics, fracture site, presence of penetrating TBI, presence of subarachnoid haemorrhage, associated neurosurgical procedures (craniotomy, cranioplasty), neurologic and functional assessments, brain imaging, occurrence of seizure, presence and type of anticonvulsant therapy, death during hospitalization.

The investigator analysed through logistic regression variables predictors of risk occurrence of seizure, and neurological and functional outcome, respectively assessed with the Glasgow Coma Scale (GCS) and the Functional Independence Measure (FIM).

DETAILED DESCRIPTION:
Seizures represent a well-known complication of acute brain injury (ABI). They can occur from the first days up to several years after ABI, with different pathophysiological mechanisms mainly depending on when they occur. In particular, acute symptomatic seizures , which occur within seven days from ABI, are thought to be directly related to acute and possibly reversible neuronal dysfunction, whereas unprovoked seizures (US), which occur after more than seven days, might follow structural changes in neuronal networks. US are associated with a persistent predisposition to generate seizures, being therefore part of an epilepsy condition. Treatment of US with antiepileptic drugs (AEDs) soon after their first appearance represents the standard care after ABI, regardless of their etiology. Beyond this practice, the post-ABI indiscriminate prescription of AEDs as preventive therapy for seizures remains controversial, even though they can potentially affect neurological outcomes in many conditions, such as TBI, ischemic and hemorrhagic stroke, and in ABI patients undergoing craniectomy or craniotomy. As a major concern, the use of AEDs for seizure prophylaxis seems to be irrelevant for the neurological outcome and mortality, and to increase the frequency of side effects, such as cognitive and behavioral complications. In this multicentric italian study, we conducted a prospective analysis on the occurrence of seizures and use of AEDs in a large cohort of patients with ABI admitted to rehabilitation, evaluating data available from admission to up to 6 months after TBI. The aim was to evaluate the effects of newly occurring seizures and of AED therapy on functional outcome, and the efficacy of AEDs as preventive treatment for seizures.

The inclusion criteria were the following: 1) age ≥ 18; 2) diagnosis of TBI on presentation; 3) admission to a hospital emergency department within 24 h of injury; 4) admission within one month from the injury to the rehabilitation unit to continue clinical care and rehabilitation program; 5) up to 6 months of observation in rehabilitation setting.

Were collected the following variables: gender, medical history, age at occurrence of injury, injury characteristics, fracture site, presence of penetrating TBI, presence of subarachnoid haemorrhage, associated neurosurgical procedures (craniotomy, cranioplasty), neurologic and functional assessments, brain imaging, occurrence of seizure, presence and type of anticonvulsant therapy, death during hospitalization. Furthermore, were specifically recorded the occurrence of seizures during both acute and rehabilitation hospitalizations. Finally, were collected data from the Glasgow Coma Scale (GCS) and the Functional Independence Measure (FIM), respectively to evaluate the neurological and functional outcome. GCS is used not only to classify severity of TBI and trend its course, but also as a validated predictor of clinical outcome after TBI.

The investigator analysed through logistic regression variables predictors of risk occurrence of seizure, and neurological and functional outcome, respectively assessed with the GCS and the FIM.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years;
* diagnosis of Traumatic Brain injury;
* admission to our rehabilitation unit within one month from the brain injury to continue clinical care and rehabilitation programs started in the intensive care unit (ICU);
* at least 6 months of observation before the discharge.

Exclusion Criteria:

* previous brain injury, or any other neurological disease;
* history of epilepsy and/or concurrent use of AEDs;
* AED prescription for psychiatric disorders;
* lack of detailed clinical data about the care during the acute phase.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this multicentric italian prospective study were enrolled adult patients admitted to intesive inpatients rehabilitation programme afther traumatic brain injury.
  The following data were collected: age at the time of the brain injury, sex, presence of subarachnoid hemorrhage, associated neurosurgical procedures, neurological and functional assessments, occurrence of seizures in either the intensive care or rehabilitation units, use and type of AEDs, death during hospitalization.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
seizure and rehabilitation | 1 years
  The predictive role of post-traumatic seizure on rehabilitation outcome, assessed with the Functional Independence Measure (FIM).
  The FIM is an 18-item measurement tool that explores a person's disability in terms of burden of care. Each of the 18 items is graded on a scale of 1-7 based on level of independence (1 = total assistance required, 7 = complete independence). The possible total score ranges from 18 (lowest) to 126 (highest) level of independence.

SECONDARY OUTCOMES:
antiepileptic drugs and rehabilitation | 1 years
  The predictive role of antiepileptic prophylactic therapy on rehabilitation outcome, assessed with the Functional Independence Measure (FIM).
  The FIM is an 18-item measurement tool that explores a person's disability in terms of burden of care. Each of the 18 items is graded on a scale of 1-7 based on level of independence (1 = total assistance required, 7 = complete independence). The possible total score ranges from 18 (lowest) to 126 (highest) level of independence.

CONTACTS AND LOCATIONS:
Locations (1):
- ICS Maugeri, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pease M, Mittal A, Merkaj S, Okonkwo DO, Gonzalez-Martinez JA, Elmer J, Liou WS, Pingue V, Hammond FM, Abramovici S, Castellano J, Barot N. Early Seizure Prophylaxis in Mild and Moderate Traumatic Brain Injury: A Systematic Review and Meta-Analysis. JAMA Neurol. 2024 May 1;81(5):507-514. doi: 10.1001/jamaneurol.2024.0689. PMID 38587858